CLINICAL TRIAL: NCT04041466
Title: Validation of the Watch Withings HWA08 for the Detection of Atrial Fibrillation
Brief Title: Validation Study of a Watch for the Detection of Atrial Fibrillation
Acronym: MOVE-ECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Withings (Industry)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A00721-56
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation; Arrythmia, Cardiac
Keywords: Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular diseases; Heart diseases; Wearable Electronic Devices; Electrocardiography
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atrial fibrillation (AF) (Experimental): Patients diagnosed with AF during reference ECG
  Interventions: Diagnostic Test: AF detection by ECG
- Sinus Rhythm (SR) (Experimental): Patients diagnosed with SR during reference ECG
  Interventions: Diagnostic Test: AF detection by ECG
- Other Arrythmia (Experimental): Patients diagnosed with an arrhythmia other than AF during the reference ECG
  Interventions: Diagnostic Test: AF detection by ECG

INTERVENTIONS:
Diagnostic Test: AF detection by ECG — Single-lead ECG with Withings watch HWA08 and reference 12-lead ECG

SUMMARY:
The proposed clinical study aims at validating the diagnostic performance, in comparison with a reference ECG, of Withings HWA08 watch for the automatic identification of atrial fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

* adults, men or women, at least 18 years old
* person having signed the informed consent form
* person affiliated to a social security system

Exclusion Criteria:

* vulnerable subject according to current regulation:

  * pregnant woman, parturient or breastfeeding
  * subject deprived of freedom by judicial, medical or administrative decision
  * subject legally protected or unable to express his consent
  * subject non-beneficiary of healthcare
  * subject falling into more than one of the above categories
* subject who refused to participate in the study
* subject in linguistic or psychic incapacity to sign a written informed consent form
* subject in physical incapacity to wear a watch on their wrist
* subject with electrical stimulation by pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
AF and SR classification accuracy | 1 visit (30 minutes)
  sensitivity and specificity of detection of AF and SR from 1-lead ECG against reference 12-lead ECG

SECONDARY OUTCOMES:
Quality of the 1-lead ECG strips | 1 visit (30 minutes)
  sensitivity and specificity of detection of AF and SR from 1-lead ECG strips reviewed by a blind, trained cardiologist against reference 12-lead ECG
safety evaluation | 1 visit (30 minutes)
  frequency of adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique AXIUM Centre de cardiologie, Aix-en-Provence
  - Centre Cardiologique du Nord, Saint-Denis

IPD SHARING:
Plan to Share IPD: No